CLINICAL TRIAL: NCT00765518
Title: Intramyocardial Delivery of Autologous Bone Marrow Cells in Patients With Heart Failure Due to Dilated Cardiomyopathy
Brief Title: Use of Ixmyelocel-T (Formerly Cardiac Repair Cell [CRC] Treatment) in Patients With Heart Failure Due to Dilated Cardiomyopathy (IMPACT-DCM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vericel Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABI-55-0712-1
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Dilated Cardiomyopathy
Keywords: Ischemic Dilated Cardiomyopathy; Non-Ischemic Dilated Cardiomyopathy; ixmyelocel-T
MeSH Terms: conditions — Cardiomyopathy, Dilated | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ixmyelocel-T (Experimental): The treatment arm of the study will receive injections of the study cellular product.
  Interventions: Biological: Ixmyelocel-T
- Standard of Care (Other): Standard of care therapy only.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Biological: Ixmyelocel-T — CRCs will be administered via direct injection into the heart muscle.
  Arms: Ixmyelocel-T
Other: Standard of Care — Because the eligible patients had no other cardiac surgery or percutaneous cardiac interventions that were likely to produce clinical improvement, SOC was limited to pharmacologic therapy, heart transplant, or ventricular assist device therapy.
  Arms: Standard of Care

SUMMARY:
This study is designed to assess the safety and tolerability of Cardiac Repair Cells (CRCs) compared to standard-of-care in patients with dilated cardiomyopathy (DCM).

DETAILED DESCRIPTION:
Heart failure remains a major public health problem, affecting 5 million patients in the US with 550,000 new diagnoses made each year. Heart failure is the leading cause of hospitalization in persons over 65 years of age with cost exceeding $29 billion annually. Prognosis is very poor once a patient has been hospitalized with heart failure. The mortality risk after heart failure hospitalization is 11.3% at 30 days, 33.1% at 1 year and well over 50% within 5 years (Hunt SA; et al., 2005). These numbers emphasize the need to develop and implement more effective treatments to manage heart failure.

This study is targeting a subset of heart failure patient population, namely those diagnosed with dilated cardiomyopathy (DCM). The World Health Organization (WHO) defines dilated cardiomyopathy as a cardiac condition wherein a ventricular chamber exhibits increased diastolic and systolic volume and a low (<40%) ejection fraction. DCM is reported to affect 108,000 to 150,000 patients in the U.S.

This study is a prospective, stratified, randomized, open-label, controlled, multi-center study to assess the safety profile and efficacy of CRCs in treating patients with DCM. It will enroll a total of 40 patients at 5 sites in the U.S.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ischemic or nonischemic DCM according to World Health Organization criteria; OR ischemic DCM (DCM in a patient with a history of myocardial infarction or evidence of clinically significant (>/= 70% narrowing of a major epicardial artery) coronary artery disease)
* No other cardiac surgery or percutaneous cardiac interventions likely to produce clinical improvement, in the opinion of the investigator and the referring interventional cardiologist
* Left ventricular ejection fraction </= 30% by echocardiogram
* Symptomatic heart failure in NYHA functional class III or IV
* Able to comply with scheduled visits in cardiac out-patient clinic
* Able to tolerate study procedures, including bone marrow aspiration, left lateral thoracotomy or thoracoscopy with single lung ventilation, MRI or cardiac CT, spirometry and 6 minute walk test
* Males and females, 18-86 years of age
* Life expectancy of 6 months or more in the opinion of investigator
* Able to give informed consent
* Normal organ and marrow function (Leukocytes >/= 3,000/microgram, Absolute neutrophil count >/= 1,500/microgram, Platelets >/= 140,000/microgram, AST (SGOT)/ALT (SGPT) </= 2.5 x institutional standards range) and Creatinine </= 2.5 mg/dL)
* Adequate pulmonary function (forced expiratory volume in one second [FEV1] > 50% predicted)
* Controlled blood pressure (systolic blood pressure </= 140; diastolic blood pressure </= 90 mmHg) and established anti-hypertensive therapy as necessary prior to entry into the study
* Adequate medical management of DCM and other pre-existing conditions. Drug treatment regimen must have been established for at least a month prior to randomization in eligible patients.
* Fertile patients must agree to use an appropriate form of contraception while participating in the study

Exclusion Criteria:

* Severe primary valvular insufficiency(ies)
* Known history of Chronic Obtrusive Pulmonary Disease (Gold stages IIB or more severe only) or restrictive pulmonary disease
* Known history of primary pulmonary hypertension
* Ventricular Assist Device implantation
* Myocardial infarction within 4 weeks of randomization
* Life-threatening ventricular arrhythmia, except if implantable cardioverter defibrillator is implanted
* Unstable angina, characterized by increasingly frequent episodes with modest exertion or at rest, worsening severity, and prolonged duration
* Patients receiving treatment with hematopoietic growth factors
* Patients who require uninterruptible anticoagulation or anti-platelet therapy [i.e. anticoagulation therapy (e.g. warfarin) that cannot be stopped for 72 hours prior to bone marrow aspiration and intramyocardial injections]
* Patients receiving anti-platelet therapy (e.g. clopidogrel) that cannot be stopped for 7 days prior to bone marrow aspiration and intramyocardial injections
* Known cancer and undergoing treatment including chemotherapy and radiotherapy
* Patients who will require continuous, systemic, high dose corticosteroid therapy (more than 7.5 mg/day) within 6 months after surgery
* End stage renal disease requiring dialysis
* Patients pregnant or lactating; positive for hCG
* History of alcohol consumption regularly exceeding the equivalent of 2 drinks/day (1 drink = 5 oz of wine or 12 oz [360mL] of beer or 1.5 oz [45mL] of hard liquor) or history of illicit drug use within 6 months of screening
* Known allergies to protein products (horse or bovine serum, or porcine trypsin)
* Body Mass Index of 40 Kg/m2 or greater
* Patients receiving experimental medications or participating in another clinical study within 30 days of screening
* HIV or syphilis, positive at time of screening
* Active Hepatitis B, or Hepatitis C infection at time of screening
* In the opinion of the investigator, patient is unsuitable for cellular therapy
* Patients receiving anti-angiogenic drugs

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-09; Primary Completion 2012-09-05 (Actual); Study Completion 2012-09-05 (Actual)

PRIMARY OUTCOMES:
Safety will be assessed by: post-procedure assessments, physical exam, vital signs, laboratory tests, and adverse events including MACE (Major Adverse Cardiac Event) occurrences. | Outcome measures will generally be assessed at baseline, Month 1, Month 3, Month 6 and Month 12

SECONDARY OUTCOMES:
Efficacy will be assessed by: MACE, myocardial size, function and perfusion; exercise tolerance, pulmonary function, medication usage, functional status, quality of life, surgical interventions, and blood markers for heart failure | Outcome measures will generally be assessed at baseline, Month 1, Month 3, Month 6 and Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Amit Patel, MD, Principal Investigator — University of Utah
Locations (5):
- United States (5):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Cleveland Clinic Heart and Vascular Institute, Cleveland, Ohio
  - Baylor University Medical Center, Dallas, Texas
  - Methodist DeBakey Heart & Vascular Center, Houston, Texas
  - The University of Utah School of Medicine, Salt Lake City, Utah

REFERENCES:
- [Derived] Henry TD, Traverse JH, Hammon BL, East CA, Bruckner B, Remmers AE, Recker D, Bull DA, Patel AN. Safety and efficacy of ixmyelocel-T: an expanded, autologous multi-cellular therapy, in dilated cardiomyopathy. Circ Res. 2014 Sep 26;115(8):730-7. doi: 10.1161/CIRCRESAHA.115.304554. Epub 2014 Aug 20. PMID 25142002